CLINICAL TRIAL: NCT05131191
Title: Application of New Algorithm ISR-Net in Measuring CT-FFR of Coronary In-stent Stenosis.
Brief Title: CT-FFR for Coronary In-stent Stenosis Based on ISR-Net Algorithm
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Xue Yu, project manager, Beijing Hospital
Other Study IDs: CT-FFR for in-stent lesion
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Coronary Stent Occlusion
Keywords: in-stent stenosis; CT derived fractional flow reserve; artificial intelligence; deep learning; image processing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with coronary metal stents implantation
  Interventions: Diagnostic Test: CT-FFR measurement; Procedure: invasive FFR

INTERVENTIONS:
Diagnostic Test: CT-FFR measurement — Patients were scanned with ≥ 64 row CT according to standard operating specifications. The software obtains the coronary CT angiography image file through the data communication interface. Based on the image processing algorithm, the centerline and contour of the target vessel can be extracted, and then the target vessel can be reconstructed to obtain the three-dimensional size information of the vessel; Based on hydrodynamics calculation and analysis, the fractional flow reserve (FFR) of each position of the target vessel is measured.
  Other Names: FFRCT
Procedure: invasive FFR — Insert the pressure guide wire into the finger guide tube and push the pressure guide wire until the pressure sensor just comes out of the orifice of guiding catheter; Equalize PD and PA values;Push the pressure guide wire to the distal end of the lesion, and record the measured blood vessel and position;Record the resting Pd / PA of the pressure guide wire;Nitroglycerin and adenosine triphosphate were administered intravenously according to standard catheter laboratory specifications to achieve maximum hyperemia;Record the FFR value of the in-stent lesions.
  Other Names: pressure wire

SUMMARY:
CT-FFR(CT-derived flow reserve fraction) usually could not been measured accurately for in-stent lesions due to the serious interference with the metal structs. ISR-Net is a new algorithm in assessing the flow of coronary in-stent stenosis. We compare the CT-FFR value of in-stent lesions with the invasive FFR measured by pressure wire to evaluate the accuracy of ISR-Net algorithm. The research results are of great significance to solve the bottleneck problem of CT-FFR and expand its application scope.

DETAILED DESCRIPTION:
CT-FFR is an important noninvasive examination to evaluate the function of coronary artery disease. It can help clinicians make clinical decisions and reduce patients' invasive coronary angiography (ICA). The image quality of coronary CT angiography (CCTA) is the basis of CT-FFR measurement. Because metal stents seriously interfere with the imaging of CCTA, it is very difficult to measure the CT-FFR value of lesions in stents. However, a large number of patients need imaging follow-up evaluation after stenting. In the previous research, the investigators creatively invented a new algorithm ISR-Net and conducted a retrospective analysis. It is preliminarily proved that the algorithm can more accurately display the stenosis lesions in the stent than the previous imaging software, making it possible to calculate the CT-FFR of the lesions in the stent. At present, the algorithm has applied for a national invention patent. In order to transform to clinical application, further clinical verification is needed. This study will evaluate the accuracy of ISR-Net algorithm in assessing the function of coronary stent stenosis by carrying out prospective clinical trials and taking the blood flow reserve fraction (FFR) measured by pressure wire as the gold standard. At the same time, the standard process of CT-FFR measurement of in stent lesions was established. The research results are of great significance to solve the bottleneck problem of CT-FFR and expand its application scope.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Over 18 years old;
* Be able to understand the purpose of the test and sign the informed consent form;
* Previous intracoronary stent implantation;
* According to the comprehensive clinical evaluation, coronary angiography and FFR were proposed;

CTA image Inclusion Criteria:

* The coronary CT angiography images showed that the reference vessel diameter of the stenosis segment in the stent was ≥ 2mm;
* The stenosis degree of coronary stent diameter ≥ 30% and ≤ 90% by visual inspection.

Exclusion Criteria:

General exclusion criteria:

* Previous coronary artery bypass grafting (CABG), artificial heart valve implantation, pacemaker or implantable defibrillator implantation;
* There are persistent or active symptoms of clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure state (systolic blood pressure less than 90 mmHg), severe congestive heart failure (NYHA cardiac function grade III or IV) or acute pulmonary edema;
* Acute myocardial infarction occurred within 7 days before enrollment;
* Patients with other severe diseases are not suitable for clinical trials, such as complex congenital heart history, sick sinus syndrome, long QT syndrome, severe arrhythmia or tachycardia, severe asthma, severe or very severe chronic obstructive pulmonary disease, chronic renal function impairment (serum creatinine value > 1.5 mg / dL or creatinine clearance rate < 45ml / kg · 1.73m2);
* There are contraindications to the use of disodium adenosine triphosphate;
* Allergic to iodized contrast media;
* Pregnancy or unknown pregnancy status;
* The expected life is less than 2 months;
* There are any other factors that the researchers believe are not suitable for inclusion or completion of this study.

CTA image exclusion criteria:

* The coronary artery image was obviously misplaced;
* Coronary artery occlusion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were implanted metal stents previously and had indications for coronary CTA test. The CT-FFR for in-stent lesions were evaluated based on Coronary CTA. Patients had the indication for invasive coronary angiography would be admitted in Cath lab and perform FFR measurement with pressure wire .
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
To predict the sensitivity, specificity and accuracy of CT-FFR in the functional sense of in stent lesions based on ISR-Net algorithm. | one month

SECONDARY OUTCOMES:
To predict the functional accuracy of in stent lesions, PPV, NPV and area under ROC curve (AUC) | one month

CONTACTS AND LOCATIONS:
Overall Officials: Xue Yu, MD, Study Chair — Beijing Hospital, National Center of Gerontology
Locations (1):
- Beijing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Z, Zhang J, Xu L, Yang W, Li G, Ding D, Chang Y, Yu M, Kitslaar P, Zhang S, Reiber JHC, Arbab-Zadeh A, Yan F, Tu S. Diagnostic Accuracy of a Fast Computational Approach to Derive Fractional Flow Reserve From Coronary CT Angiography. JACC Cardiovasc Imaging. 2020 Jan;13(1 Pt 1):172-175. doi: 10.1016/j.jcmg.2019.08.003. Epub 2019 Sep 18. No abstract available. PMID 31542542
- [Background] Tang CX, Liu CY, Lu MJ, Schoepf UJ, Tesche C, Bayer RR 2nd, Hudson HT Jr, Zhang XL, Li JH, Wang YN, Zhou CS, Zhang JY, Yu MM, Hou Y, Zheng MW, Zhang B, Zhang DM, Yi Y, Ren Y, Li CW, Zhao X, Lu GM, Hu XH, Xu L, Zhang LJ. CT FFR for Ischemia-Specific CAD With a New Computational Fluid Dynamics Algorithm: A Chinese Multicenter Study. JACC Cardiovasc Imaging. 2020 Apr;13(4):980-990. doi: 10.1016/j.jcmg.2019.06.018. Epub 2019 Aug 14. PMID 31422138
- [Background] Coenen A, Kim YH, Kruk M, Tesche C, De Geer J, Kurata A, Lubbers ML, Daemen J, Itu L, Rapaka S, Sharma P, Schwemmer C, Persson A, Schoepf UJ, Kepka C, Hyun Yang D, Nieman K. Diagnostic Accuracy of a Machine-Learning Approach to Coronary Computed Tomographic Angiography-Based Fractional Flow Reserve: Result From the MACHINE Consortium. Circ Cardiovasc Imaging. 2018 Jun;11(6):e007217. doi: 10.1161/CIRCIMAGING.117.007217. PMID 29914866
- [Background] Ko BS, Cameron JD, Munnur RK, Wong DTL, Fujisawa Y, Sakaguchi T, Hirohata K, Hislop-Jambrich J, Fujimoto S, Takamura K, Crossett M, Leung M, Kuganesan A, Malaiapan Y, Nasis A, Troupis J, Meredith IT, Seneviratne SK. Noninvasive CT-Derived FFR Based on Structural and Fluid Analysis: A Comparison With Invasive FFR for Detection of Functionally Significant Stenosis. JACC Cardiovasc Imaging. 2017 Jun;10(6):663-673. doi: 10.1016/j.jcmg.2016.07.005. Epub 2016 Oct 19. PMID 27771399
- [Background] Coenen A, Lubbers MM, Kurata A, Kono A, Dedic A, Chelu RG, Dijkshoorn ML, van Geuns RJ, Schoebinger M, Itu L, Sharma P, Nieman K. Coronary CT angiography derived fractional flow reserve: Methodology and evaluation of a point of care algorithm. J Cardiovasc Comput Tomogr. 2016 Mar-Apr;10(2):105-13. doi: 10.1016/j.jcct.2015.12.006. Epub 2015 Dec 18. PMID 26747231
- [Background] Fuchs A, Kuhl JT, Chen MY, Helqvist S, Razeto M, Arakita K, Steveson C, Arai AE, Kofoed KF. Feasibility of coronary calcium and stent image subtraction using 320-detector row CT angiography. J Cardiovasc Comput Tomogr. 2015 Sep-Oct;9(5):393-8. doi: 10.1016/j.jcct.2015.03.016. Epub 2015 Apr 16. PMID 26091841